CLINICAL TRIAL: NCT01536301
Title: Evaluation of Oxycodone Hydrochloride Versus Intravenous Morphine Hydrochloride for Postoperative Analgesia After Hip Prosthetic Surgery
Brief Title: Oxycodone Versus Intravenous Morphine for Postoperative Analgesia After Hip Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LOCAL/2011/PC-02; 2011-004140-22 (EudraCT Number)
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2018-01

CONDITIONS: Arthroplasty, Replacement, Hip
Keywords: oxycodone; morphine; hip replacement; analgesia; post operative analgesia
MeSH Terms: conditions — Agnosia | interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Morphine (Active Comparator): The patients in this arm will have post-operative analgesia including morphine (patient controlled analgesia).
  Interventions: Drug: Standard Care morphine hydrochloride
- Oxycodone (Experimental): The patients in this arm will have post operative analgesia including oxycodone (patient controlled analgesia).
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Standard Care morphine hydrochloride — Post-operative analgesia including morphine (patient controlled analgesia).
  Other Names: morphine hydrochloride
  Arms: Morphine
Drug: Oxycodone — Post-operative analgesia including oxycodone (patient controlled analgesia).
  Other Names: oxycodone hydrochloride
  Arms: Oxycodone

SUMMARY:
The main objective is to demonstrate that postoperative analgesia by IV oxycodone (compared to morphine IV) reduces opioid-related adverse events (nausea, vomiting, pruritus, respiratory depression, urinary retention, allergies, hallucination) by 50% in adult patients operated on for prosthetic hip surgery.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for a 4 month follow-up
* The patient weight between 50 and 100 kg
* Patient scheduled for unilateral hip arthroplasty
* Patient has creatinine clearance > 50 ml/min (Cockroft)
* Patient with ASA-PS score of 1, 2 or 3 (American Society Anesthesiology - Physical Status)

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* Patient with ASA score of 4
* Patient has a known deficit in cytochrome P450
* Uncontrolled epilepsy
* Chronic alcoholism
* Patient already taking opiate agonist on a long term basis (codeine, dextromoramide, dihydrocodeine, oxycodone po, morphine-like antitussif)
* Patient already taking agonist-antagonists on a long term basis (buprenorphine, nalbuphine, pentazocine)
* The patient is under treatment for liver inducing enzyme cytochrome P450: anti-infectives (e.g. rifampicin, rifabutin, nevirapine, griseofulvin), antiepileptic (phenobarbital, phenytoin)
* the patient has an allergy to opiates
* the patient has chronic renal insufficiency: creatinine clearance < 50 ml / min (Cockroft formula)
* the patient has severe hepatic insufficiency(transaminase and/or alkaline phosphatase x 3/nal))
* patient with porphyria, intracranial hypertension, a syndrome subocclusive or ileus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2012-06; Primary Completion 2016-11-15 (Actual); Study Completion 2016-11-15 (Actual)

PRIMARY OUTCOMES:
Composite score of complications | 24 hours
  The presence/absence of at least one of the following complications: nausea, vomiting, respiratory depression, pruritus (itch), urinary retention requiring evacuation (spontaneous voiding impossible despite bladder volume> 400 ml measured by ultrasound), allergy (skin reaction, hallucination (perception without object).
  Drowsiness (Ramsay score) is not considered an adverse event within the primary endpoint.

SECONDARY OUTCOMES:
Number of opioid boluses in the post-intervention surveillance room | Day 1
Time to obtain a VAS score < 30/100 (from the first administration; minutes) | Day 1
Length of stay in the post-intervention surveillance room (minutes) | Day 1
Total dose of opioids during the first 24 hours (mg) | 24 hours
Total number of opioid requestions (patient controlled analgesia = PCA) | Day 1
Total number of opioid requestions (patient controlled analgesia = PCA) | Day 2
Total number of opioid requestions (patient controlled analgesia = PCA) | Day 3
Total number of opioid requestions accepted / refused (PCA) | Day 1
Total number of opioid requestions accepted / refused (PCA) | Day 2
Total number of opioid requestions accepted / refused (PCA) | Day 3
Ramsay score | Day 1
Ramsay score | Day 2
Ramsay score | Day 3
Presence / absence of an overdose of morphine/oxycodone (Ramsay score > 4) | Day 1
Presence / absence of an overdose of morphine/oxycodone (Ramsay score> 4) | Day 2
Presence / absence of an overdose of morphine/oxycodone (Ramsay score> 4) | Day 3
Presence/absence of complications | Day 1
  nausea, vomiting, respiratory depression, pruritus, urinary retention, allergy to morphine or oxycodone, hallucinations, psychiatric disorders, constipation
Presence/absence of complications | Day 2
  nausea, vomiting, respiratory depression, pruritus, urinary retention, allergy to morphine or oxycodone, hallucinations, psychiatric disorders, constipation
Presence/absence of complications | Day 3
  nausea, vomiting, respiratory depression, pruritus, urinary retention, allergy to morphine or oxycodone, hallucinations, psychiatric disorders, constipation
Patient satisfaction, VAS scale | Hospital discharge
Patient satisfaction, VAS scale | 4 months
Pain while at rest at while moving (Visual Analog Scale) | Day -1 (before intervention)
Pain while at rest at while moving (Visual Analog Scale) | Day 1
Pain while at rest at while moving (Visual Analog Scale) | Day 2
Pain while at rest at while moving (Visual Analog Scale) | Day 3
DN4 score | Day -1 (before intervention)
DN4 score | 4 months
Length of hospital stay (hours) | Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Lana Zoric, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes; Philippe Cuvillon, MD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, Gard
  - APHP - Groupe Hospitalier Pitié-Salpetrière, Paris

REFERENCES:
- [Result] Cuvillon P, Alonso S, L'Hermite J, Reubrecht V, Zoric L, Vialles N, Luc Faillie J, Kouyoumdjian P, Boisson C, Raux M, Langeron O. Post-operative opioid-related adverse events with intravenous oxycodone compared to morphine: A randomized controlled trial. Acta Anaesthesiol Scand. 2021 Jan;65(1):40-46. doi: 10.1111/aas.13685. Epub 2020 Sep 27. PMID 32790073